CLINICAL TRIAL: NCT07009041
Title: The Effects Of An Integrated Training Program On Jump Performance And Knee Valgus In Youth Football Players: A Controlled Group Study
Brief Title: Integrated Training Program On Jump Performance And Knee Valgus In Youth Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Vesile Şahiner Güler, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERU-SAGENS-VSG-01
Record Dates: First submitted 2025-05-14; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Knee Valgus
Keywords: Football; jump performance; anterior cruciate ligament; knee valgus; injury prevention; exercise training program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The group that received 8-week training programs
  Interventions: Other: Strength training program; Other: Stretching exercises program; Other: Plyometric exercises program; Diagnostic Test: Demographic tests; Diagnostic Test: Jump tests; Diagnostic Test: Knee Valgus tests
- Control Group (Other): Group without any intervention
  Interventions: Diagnostic Test: Demographic tests; Diagnostic Test: Jump tests; Diagnostic Test: Knee Valgus tests

INTERVENTIONS:
Other: Strength training program — Strength training was implemented for eight weeks, including full-body, core, and leg exercises.
  Arms: Experimental Group
Other: Stretching exercises program — Stretching exercises were performed after strength training for the entire eight-week period. The training was administered exclusively to participants in the experimental group, following a consistent schedule and sequence. The program was conducted three days a week for eight weeks, separate from regular football training.
  Arms: Experimental Group
Other: Plyometric exercises program — Plyometric exercises were included only one day per week, and a minimum one-day rest period was maintained between training sessions.Since this program was originally 6 weeks long, it was implemented in the first 6 weeks of the study's implementation process.
  Arms: Experimental Group
Diagnostic Test: Demographic tests — Demographic tests were applied to determine the height, weight and BMI values for the identification of the participants.
Diagnostic Test: Jump tests — Jump tests (CMJ, CMJ Free, SJ, DJ, Horizontal Jump). Three different measurements were taken at three different times.(Before starting, end of week 4 and after completion of week 8).
Diagnostic Test: Knee Valgus tests — It was conducted to determine the right and left knee valgus values of the participants.Three different measurements were taken at three different times. (Before starting, end of week 4 and after completion of week 8).

SUMMARY:
This study aimed to investigate the effects of stretching, strength, and plyometric exercise training programs, applied in addition to regular training, on jumping performance and knee valgus values in football players.

DETAILED DESCRIPTION:
The sample of this study consisted of male football players from an under-19 (U-19) team based in Kayseri, Turkey. The inclusion criteria required participants to be male, aged 18 or older, actively competing in the U-19 category, free from any disabilities, and to have at least five years of experience as licensed football players. In 2024, ninety athletes from an amateur football club were invited to participate in the study. Participants were assigned to experimental and control groups using an unbiased sampling method. Groups were balanced based on pre-test results to ensure equivalence.

A true experimental design was employed, specifically the pre-test-post-test control group model. Jump tests, including the countermovement jump (CMJ), free-arm countermovement jump (CMJFREE), drop jump (DJ), squat jump (SJ), and horizontal jump, were conducted using the My Jump 2 application. The knee valgus test was performed using the My Jump Lab application, which enables markerless motion analysis by evaluating images recorded by a mobile device. This application provides valuable insights into injury prevention particularly in the lower extremities and supports the assessment of proper execution of technical movements.

The training program included strength, flexibility, and plyometric exercises, designed to reduce muscle strength imbalances while enhancing flexibility and plyometric performance. Since improvements in motor characteristics and muscle balance are expected to positively affect knee valgus angles, all components of the training program were implemented in combination. Strength training was carried out over eight weeks and included full-body, core, and lower extremity exercises. In addition, the anterior cruciate ligament injury prevention program developed by Hewett et al., which emphasizes plyometric training, was incorporated during the first six weeks in accordance with its prescribed duration. Stretching exercises were performed following strength training sessions throughout the entire eight-week period. The training program was administered exclusively to the experimental group and followed a consistent schedule and sequence. Training sessions were conducted three times per week for eight weeks, separate from routine football practices. Plyometric exercises were included once per week, and a minimum one-day rest interval was maintained between sessions.

Data were analyzed using SPSS version 27. The Kolmogorov-Smirnov test was used to assess the normality of data distribution. Repeated Measures Analysis of Variance (ANOVA) was applied for within-subject comparisons, while the Bonferroni test was used to determine the source of significant differences. Between-group comparisons were conducted using the Independent Samples t-test.

ELIGIBILITY:
Inclusion Criteria:

* Being a football player playing in the U-19 football team
* Being a male
* Residing in Kayseri
* Be between 18-19 years old

Exclusion Criteria:

* Not being a football player playing on the U-19 football team
* Being a female
* Residence outside Kayseri
* Being outside the 18-19 age range

Ages: 18 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 90 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Change in Countermovement Jump Height (CMJ) Measured in Centimeters | Each participant in the study was evaluated by taking 3 separate measurements before starting the study, at the end of the 4th week of the study, and at the end of the 8th week of the study. The total evaluation process was completed within 8 weeks.
  CMJ test was performed using the My Jump 2 app. The jump height (in cm) was recorded in 3 separate measurements and the average was used for comparison.Unit of Measure: Centimeters (cm)
Change in Free Arm Countermovement Jump Height (CMJFREE) Measured in Centimeters | Each participant in the study was evaluated by taking 3 separate measurements before starting the study, at the end of the 4th week of the study, and at the end of the 8th week of the study. The total evaluation process was completed within 8 weeks.
  CMJFREE test was performed using the My Jump 2 app with free arm movement. Values were averaged from 3 trials.Unit of Measure: Centimeters (cm)
Change in Drop Jump Height (DJ) Measured in Centimeters | Each participant in the study was evaluated by taking 3 separate measurements before starting the study, at the end of the 4th week of the study, and at the end of the 8th week of the study. The total evaluation process was completed within 8 weeks.
  DJ test was performed using the My Jump 2 app. Jump height (cm) was measured and averaged across 3 attempts.Unit of Measure: Centimeters (cm).
Change in Squat Jump Height (SJ) Measured in Centimeters | Each participant in the study was evaluated by taking 3 separate measurements before starting the study, at the end of the 4th week of the study, and at the end of the 8th week of the study. The total evaluation process was completed within 8 weeks.
  SJ test was performed using the My Jump 2 app. Jump height (cm) was measured and averaged across 3 trials.Unit of Measure: Centimeters (cm)
Change in Horizontal Jump Distance Measured in Centimeters | Each participant in the study was evaluated by taking 3 separate measurements before starting the study, at the end of the 4th week of the study, and at the end of the 8th week of the study. The total evaluation process was completed within 8 weeks.
  Horizontal jump test was performed manually. Jump distance (cm) was recorded and averaged across 3 trials.Unit of Measure: Centimeters (cm)
Change in Knee Valgus Angle Measured in Degrees | Each participant in the study was evaluated by taking 3 separate measurements before starting the study, at the end of the 4th week of the study, and at the end of the 8th week of the study. The total evaluation process was completed within 8 weeks.
  Knee valgus angle was assessed using the My Jump Lab app. Degree values were measured from 3 trials and averaged for each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Talas, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided